CLINICAL TRIAL: NCT03971110
Title: A Multi-centre, Single-arm, Prospective Study to Assess Efficacy and Safety of Neoadjuvant Hormone Therapy Using Zoladex (Goserelin) and Casodex (Bicalutamide) in Patients With Advanced Prostate Cancer Undergoing Radical Prostatectomy.
Brief Title: A Study of Neoadjuvant Hormone Therapy in Patient With Advanced Prostate Cancer Undergoing Radical Prostatectomy.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to the limited potential patients pool, the enrollment goal could not be achieved. After review and communication, the decision to teminate study was made.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8664C09827
Record Dates: First submitted 2019-03-21; First posted 2019-06-03 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Advanced Prostate Cancer
MeSH Terms: interventions — Goserelin; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zoladex and Casodex (Experimental): Subjects who are diagnosed with advanced prostate cancer at clinical stage of T3 and T4 (N0 or N1, M0 or M1 with five or fewer extra-pelvic lesions) are the target population of this study. The eligible subjects will receive Casodex 50 mg orally per day in combination with Zoladex 10.8 mg implant subcutaneously as neoadjuvant therapy per 12 weeks for up to 24 weeks.
  Interventions: Drug: Zoladex and Casodex

INTERVENTIONS:
Drug: Zoladex and Casodex — The eligible subjects will receive Casodex 50 mg orally per day in combination with Zoladex 10.8 mg implant subcutaneously as neoadjuvant therapy per 12 weeks for up to 24 weeks.

SUMMARY:
This is A Multi-centre, Single-arm, Prospective, Interventional Study to Assess Efficacy and Safety of Neoadjuvant Hormone Therapy using Zoladex (Goserelin) and Casodex (Bicalutamide) in Patients with Advanced Prostate Cancer Undergoing Radical Prostatectomy, to assess the efficacy by resectability rate of neoadjuvant hormone therapy (NHT) in subjects with advanced prostate cancer.

DETAILED DESCRIPTION:
Neoadjuvant hormonal treatment (NHT) for clinically localised prostate cancer consists of complete androgen blockade (CAB) preceding either radiotherapy or surgery. The rational for this approach is based on the assumption that NHT will reduce both the tumour and normal prostatic tissue volume, and induce cancer regression by the mechanism of apoptosis [1].

Most randomized clinical trials show that NHT reduces the incidence of positive surgical margins after radical prostatectomy and apparently determines tumour downstaging, however no advantage has been documented in terms of biochemical disease progression [for example, time to prostate specific antigen (PSA) increase] between treated and untreated patients [2-8]. Because of relatively low biological aggressiveness of prostatic carcinoma, many patients will need to be followed for a considerable time before drawing significant conclusions on the effects of NHT on survival [2,4,7,10]. A large sample of 393 radical prostatectomy specimens were evaluated in 3 treatment groups, which were immediate surgery, 12 weeks of NHT (Zoladex and Casodex), and 24 weeks of NHT. Patients included clinical stage B (T2a and T2b) and stage C (T3a and T3b). Systemic hormonal treatment, whether 12 weeks or 24 weeks of NHT, is able to "downstage" the primary tumour and decrease the positive margin rate before definitive localised treatment [11].

Currently treatment of patients with oligometastatic prostate cancer is undergoing dramatic changes [12]. The local treatment of the primary tumour might provide a survival benefit to men with metastatic and lymph node-positive disease. Similar observations have been made in treatment of metastatic lesions with life-prolonging, rather than palliative intent [13-17].

This study is proposed primarily to observe the efficacy and safety of 24-week NHT (Zoladex and Casodex) in patients with locally advanced or oligometastatic prostate cancer. Progression status and survival will be followed-up for up to 2 years after NHT.

This is a multi-centre, single-arm and prospective study to explore the efficacy and safety of neoadjuvant hormone therapy (NHT) for advanced prostate cancer patients undergoing radical prostatectomy (RP). A total of 104 subjects with locally advanced and oligometastatic prostate cancer at clinical stage of T3 and T4 will be enrolled at almost 20 centres in China.

The eligible subjects will receive Casodex 50 mg orally per day in combination with Zoladex 10.8 mg implant subcutaneously every 12 weeks as neoadjuvant therapy for 24 weeks, and then will be assessed for resectability of the primary tumour. The subjects will undergo a RP [RALP (robot-assisted laparoscopic prostatectomy), laparoscopic RP or RRP (radical retropubic prostatectomy)] plus eLND thereafter if the primary tumour is assessed as resectable. Surgical margin status and involvement of bilateral pelvic lymph nodes will be evaluated. Subjects will be prescribed post-surgical treatment such as continuous ADT and metastasis-directed therapy upon investigator's discretion and be followed-up for up to 2 years.

Progression free survival (PFS) and overall survival (OS) will be collected during this study.

For the subjects with unresectable primary tumour after NHT, PFS and OS will also be collected in the follow-up for up to 2 years after 24 weeks of CAB.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed within the past 12 months with T2DM according to 1999 WHO criteria
2. Men and women aged at least 18 years at screening.
3. Either not received oral anti-diabetic drugs or had been on short-term (1 month) treatment that had been discontinued 3 months before enrolment.
4. HbA1c ≥ 7.5% and ≤ 10.5% at screening and HbA1c ≥ 7.0% and ≤ 10.5% at pre-randomization visit.
5. FPG ≤ 13.3 mmol/L (≤ 240 mg/dL) .
6. BMI≥18.5 kg/m2 and ≤ 45.0 kg/m2 .
7. C-peptide ≥0.33nmol/L(≥1.0 ng/mL).
8. Able and willing to provide written informed consent and to comply with the study.

Exclusion Criteria:

1. Women who are pregnant, intending to become pregnant during the study period, currently lactating females, or women of child-bearing potential not using highly effective, medically approved birth control methods.
2. Diagnosis or history of:

   1. Acute metabolic diabetic complications such as ketoacidosis or hyperglycemic hyperosmolar state
   2. Diabetes insipidus.
3. Requirement for insulin therapy. Symptoms of poorly controlled diabetes, including but not limited to, marked polyuria and polydipsia with >10% weight loss during the 3 months before enrollment.
4. Triglycerides (fasting) > 9.3 mmol/L (> 800 mg/dL).
5. Patients with clinically apparent hepatobiliary disease, including but not limited to chronic active hepatitis and/or severe hepatic insufficiency. ALT or AST > 3x upper limit of normal (ULN), or serum total bilirubin (TB) >34.2 μmol/L (>2 mg/dL).
6. Patiens with following renal disease history or renal disease related features:

   1. History of unstable or rapidly progressing renal disease;
   2. Patients with moderate /severe renal impairment or end-stage renal disease (eGFR< 60 mL/min/1.73 m2)
   3. Urinary albumin: creatinine ratio >1800 mg/g;
   4. Serum creatinine (Cr) ≥133 μmol/L (≥1.50 mg/dL) for male subjects; Serum Cr≥124 μmol/L (≥1.40 mg/dL) for female subjects;
   5. Conditions of congenital renal glycosuria.
7. Severe uncontrolled hypertension defined as SBP ≥180 mmHg and/or BP ≥110 mmHg;Patients with SBP < 95mmHg.
8. Any of the following cardiovascular diseases within 6 months of the enrollment visit:

   1. Myocardial infarction;
   2. Cardiac surgery or revascularization (coronary artery bypass graft/percutaneous transluminal coronary angioplasty);
   3. Unstable angina;
   4. Congestive heart failure New York Heart Association Class III or IV;
   5. Transient ischemic attack or significant cerebrovascular disease.
9. History of gastrointestinal disease or surgery including Roemheld Syndrome, severe hernia, intestinal obstruction, intestinal ulcer, gastroenterostomy, enterectomy, bariatric surgery or lap-band procedure.
10. Malignancy within 5 years of the enrollment visit (with the exception of treated basal cell or treated squamous cell carcinoma).
11. Known immunocompromised status, including but not limited to, individuals who had undergone organ transplantation or acquired immunodeficiency syndrome (AIDS).
12. Any subject who, in the judgment of the investigator, was at risk for dehydration or volume depletion that might affect the interpretation of efficacy or safety data.
13. History of bone fracture secondary to diagnosed severe osteoporosis.
14. Currently unstable or serious cardiovascular, renal, hepatic, hematologic, oncologic, endocrine, psychiatric, or rheumatic diseases as judged by the Investigator.
15. Replacement or chronic systemic corticosteroid therapy, defined as any dose of systemic corticosteroid taken for >4 weeks within 3 months before enrollment visit.
16. Administration of sibutramine, phentermine, orlistat, rimonabant, benzphetamine, diethylpropion, methamphetamine, or phendimetrazine within 30 days of enrollment visit.
17. Any subject who was currently abusing alcohol or other drugs or had done so within the last 6 months
18. Donation of blood or blood products, blood transfusion, or participation in a clinical study requiring withdrawal of >400 mL of blood during the 6 weeks before the enrollment visit
19. History of hypersensitivity reaction to dapagliflozin or acarbose. Allergies or contraindication to the contents of dapagliflozin tablets or acarbose tablests.
20. Previous participation in a clinical trial with dapagliflozin.
21. Administration of any other investigational drug within 30 days of planned enrollment to this study, or within 5 half-life periods of other investigational drugs.
22. Subject is, in the judgment of the Investigator, unlikely to comply with the protocol or has any severe concurrent medical or psychological condition that may affect the interpretation of efficacy or safety data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
Resectability rate for primary tumour (the resectability will be assessed by central review using a digital rectal examination and confirmed by CT or MRI) | at 24 week
  To assess the efficacy by resectability rate of neoadjuvant hormone therapy (NHT) in subjects with advanced prostate cancer

SECONDARY OUTCOMES:
Radical prostatectomy rate | From baseline to 24 week
  Which will be derived using the number of patient who will conduct the radical prostatectomy at 24 week.
The mean PSA by the end of NHT | From baseline to 24 week
  which will be derived using the value of mean PSA by the end of NHT
Percentage of positive surgical margin for primary tumour | From baseline to 24 week
  Which will be derived using the number of positive surgical margin at 24 week
Incidence of seminal vesicle invasion | From baseline to 24 week.
  Which will be derived using the value of incidence of seminal vesicle invasion at 24 week
Percentage of pathological downstaging | From baseline to 24 week
  Which will be derived using the number of pathological downstaging at 24 week.
surgical-related variables at 12 weeks, potent rates in erectile function at 12 weeks after surgery | From 24 week to 36 week
  Which will be derived using the value of observe surgical-related variables and complications at week 36
PFS | From baseline to the end of study
  Which will be derived using the number of PFS at the end of study
AEs/SAEs | From baseline to 28 week
  To evaluate the safety of NHT using goserelin and bicalutamide
PSA change from baseline | From baseline to 24 week
  Which will be derived using the value of PSA at the baseline.
Involvement of bilateral pelvic lymph nodes | From baseline to 24 week
  Which will be derived using the value of involvement of bilateral pelvic lymph nodes at 24 week.
OS | From baseline to the end of study
  Which will be derived using the number of OS at the end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Gao, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (12):
- China (12):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shijiazhuang
  - Research Site, Ürümqi
  - Research Site, Xi'an
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] 1. Montironi R, Schulman CC. Pathological changes in prostate lesions after androgen manipulation. J Clin Pathol 1998; 51:5-12. 2. Witjes WP, Schulman CC, Debruyne FM. Preliminary results of a prospective randomized study comparing radical prostatectomy versus radical prostatectomy associated with neoadjuvant hormonal combination therapy in T2-3 N0 M0 prostatic carcinoma. Urology 1997;49(suppl):65-9. 3. Labrie F, Cusan L, Gomez JL, et al. Neoadjuvant hormonal therapy: the Canadian experience. Urology 1997;49(suppl):56-60. 4. Soloway MS, Sharifi F, Wajsman Z, et al. Random prospective study comparing radical prostatectomy alone versus radical prostatectomy preceded by androgen blockade in clinical stage B2 (T2bNxM0) prostate cancer. J Urol 1995; 154:424-8. 5. Hugosson J, Abrahamsson PA, Ahlgren G, et al. The risk of malignancy in the surgical margin at radical prostatectomy is reduced almost three-fold in patients given neoadjuvant hormone treatment. Eur Urol 1996; 29:413-16.